CLINICAL TRIAL: NCT00899119
Title: Autologous Stem Cell Harvesting for Waldenstrom's Macroglobulinemia
Brief Title: Collecting Stem Cells in Patients With Waldenstrom's Macroglobulinemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000487602; CPMC-AAAB4806
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2008-01

CONDITIONS: Lymphoma
Keywords: Waldenström macroglobulinemia
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia | interventions — Leukapheresis

INTERVENTIONS:
Procedure: leukapheresis

SUMMARY:
RATIONALE: Collecting and storing stem cells to study in the laboratory may help doctors learn more about collecting stem cells from patients who have undergone treatment for Waldenstrom's macroglobulinemia.

PURPOSE: This laboratory study is collecting stem cells from patients with Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Harvest and store adequate CD34+ stem cells from patients with Waldenstrom's macroglobulinemia (WM) for potential future use in transplantation strategies.
* Evaluate the ability to harvest stem cells after therapy for WM (e.g., fludarabine-based chemotherapy) by evaluating the number of days to adequate harvest.
* Collect aliquots of stem cells for future research analysis as part of a WM database project.

OUTLINE: Patients undergo collection of autologous stem cells beginning on day 4 or 5 and continuing until an adequate number of stem cells are collected. Cells are then cryopreserved.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Waldenstrom's macroglobulinemia (WM)
* Less than 30% lymphoplasmacytoid cells in bone marrow by histopathology
* Received prior chemotherapy for WM

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC > 2,000/mm³
* Platelet count > 50,000/mm³
* LVEF ≥ 50%
* No organ dysfunction that would preclude future transplantation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-11

PRIMARY OUTCOMES:
Number of days to adequate stem cell harvest

CONTACTS AND LOCATIONS:
Overall Officials: Gwen L. Nichols, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York, United States